CLINICAL TRIAL: NCT04349137
Title: Cause-effect Relationships Between Brain Networks and Bimanual Coordination in Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, prof. dr. Raf Meesen, Principal Investigator, Hasselt University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: RWS-SV-001
Record Dates: First submitted 2020-04-03; First posted 2020-04-16 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Healthy Aging; Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- In-phase 6Hz tACS (Experimental): Transcranial alternating current stimulation (tACS) will be administered over the right PPC and the right DLPFC in a synchronized (in-phase) manner at a frequency of 6Hz
  Interventions: Device: HD-tACS
- Anti-phase 6Hz tACS (Active Comparator): Transcranial alternating current stimulation (tACS) will be administered over the right PPC and the right DLPFC in a desynchronized (anti-phase, i.e. with a difference of 180deg) manner at a frequency of 6Hz
  Interventions: Device: HD-tACS
- Sham tACS (Sham Comparator): A sham transcranial alternating current stimulation (tACS) will be administered over the right PPC and the right DLPFC at a frequency of 6Hz using physical vibrations instead of electrical current
  Interventions: Device: sham HD-tACS

INTERVENTIONS:
Device: HD-tACS — non-invasive high-definition dual-site transcranial alternating current stimulation (HD-tACS) low intensive electrical alternating currents (2 mA peak-to-peak) are externally applied to the skull at a frequency of 6Hz to entrain endogenous neural oscillatory activity.
  Arms: Anti-phase 6Hz tACS; In-phase 6Hz tACS
Device: sham HD-tACS — sham non-invasive high-definition dual-site transcranial alternating current stimulation (HD-tACS)
  Arms: Sham tACS

SUMMARY:
In this study, high-definition dual-site transcranial alternating current stimulation (i.e., non-invasive brain stimulation) will be applied to boost the fronto-parietal network during a bimanual coordination task in healthy young and older adults. Previous studies indicated that this network is important in initial motor learning, possibly through its role in spatial working memory. Therefore, stimulation will be applied during both a pure spatial working memory test, and during a bimanual coordination task.

It is also shown that healthy older adults do not engage spatial working memory brain regions during motor learning, which is related to worse motor learning. Therefore, the investigators will investigate whether this type of stimulation can improve bimanual motor learning in healthy older adults.

DETAILED DESCRIPTION:
A single-blind, pseudo-randomised, sham-controlled within-subject design will be used. The study consists of three experimental sessions. In each session, one out of three stimulation conditions was applied: (1) in-phase stimulation; (2) anti-phase stimulation; (3) sham stimulation. The order of the three stimulation conditions over sessions will be pseudo-randomised across participants. Within each session, stimulation is applied during the performance of two tasks: a 2-back task for assessing pure spatial working memory (sWM), and a complex bimanual tracking task (BTT) for assessing bimanual skill acquisition. To minimise learning and carry-over effects over sessions, a wash-out period of 6 weeks in between sessions is used and three different variants of the BTT task (one for each session). The order of these variants was also pseudo-randomised across participants.

For assessing sWM, participants perform an adapted version of the 2-back visuospatial match-to-sample test used in Alekseichuk et al., 2016. Participants are seated on a chair, with their right hand resting on a response box. A computer screen is placed in front of the participant. On the screen, a blue 3x3 grid is drawn on a black background. Each trial consists of three events: a stimulus, a probe, and a response period. During the stimulus, two or three white dots appear somewhere in the grid for 2150ms. After a time interval of 50ms, this is followed by the appearance of the probe, consisting of one small blue dot, lasting for 300ms. During the response period (2000ms duration), the participant is requested to either press or to not press the response button, indicating whether the location of the probe matches the location of the stimulus in the previous trial or not (i.e., 2-back condition).

For familiarisation purposes, participants are first instructed what the goal of the task is. Next, they practiced a series of ten or twenty trials without stimulation.

For the experiment (i.e., task performance during stimulation), a complete set of trials is organised in five blocks, consisting of 30 trials (i.e. 150 trials per set). The five blocks are separated by 1-minute breaks. The distribution of 2-dot or 3-dot stimulus conditions in the 150-trial set was 50%-50%, presented in random order. Forty % of the trials are matched trials (i.e. 58 trials) and 60% are non-matched trials (i.e. 87 trials).

For this study, we use three fixed sets of trials, i.e. one for each session. The order of these sets over sessions will be pseudo-randomised across participants.

For assessing initial bimanual learning, we use a complex visuomotor bimanual tracking task (BTT). Participants are seated in front of a computer screen with their arms pronated on the table. Each index finger is placed in a controller. The controllers are two rotatable dials with small grooves for finger placement. By bimanually rotating the two dials, the participant can move the position of a red cursor on the display. Left and right dial rotations induced cursor movement along the ordinate and abscissa.

The goal of the BTT is to manipulate the cursors' position in order to follow a moving target dot on a straight inclined line, presented on the display, as accurately as possible. Each BTT trial starts with the appearance of the target line. At the origin of this line, in the center of the display, a red target dot is presented for 2 seconds (i.e. preparation period). Then, an auditory GO-signal indicates the start of the movement period: the target dot begins to move at a constant speed along the line towards the peripheral end of the line, which the participant has to follow by rotating the dials simultaneously. The duration of the target dot movement from center to periphery (i.e. movement period) is 5 seconds. Between trials, a time interval of 3 seconds is implemented.

There are four different task conditions that differ in relative inter-hand frequencies (1:3 vs. 3:1) and relative directionality of the rotating dials (iso-directional [ISO] vs. non-iso-directional [NON-ISO]). More specifically, in the 1:3 condition, the right index finger has to rotate the dial three times faster than the left hand, while in the 3:1 condition, this pattern is reversed. For the ISO mode, both index fingers have to rotate the dials either to the right (ISO-R) or left (ISO-L). For the NON-ISO mode, both index fingers have to rotate the dials either inward (NON-ISO-IN) or outward (NON-ISO-OUT).

To get familiar with the task, a practice block of 16 trials without stimulation is implemented. For the experiment (i.e. task performance during stimulation), there are four blocks of 36 trials, where each task condition is repeated nine times in each block. We provide 1-minute breaks between blocks. Fifteen minutes after the end of the fourth block, a retention block of 36 trials without stimulation will be added. The order of the four task conditions within each block will be randomised.

To minimize learning effects over the three sessions, we rotated the reference frame of line orientation each time with 90 degrees.

Stimulation will be delivered by two battery-driven Direct Current (DC) stimulator PLUS devices (neuroConn and Eldith GmbH, Ilmenau, Germany). Each device is connected to a center-surround rubber ring montage, suited for focal stimulation. Each montage consists of a small circular center electrode (diameter of 20 mm) and a surrounding ring electrode (inner diameter of 40 mm and outer diameter of 60 mm). The center electrodes are positioned according to the 10-20 EEG system: in the middle between AF4 and F4, which corresponds to the junction between BA9 and BA46 (i.e. right dorsolateral prefrontal cortex (DLPFC)); and P4, which corresponds to the right posterior parietal cortex (PPC). Impedance is kept below 10kOhm using a conductive paste (Ten20, Weaver and Company, CO, USA).

In-phase stimulation will consist of 6Hz stimulation over the right DLPFC and the right PPC that is synchronized (0deg phase lag between both sites), while anti-phase stimulation will use desynchronized 6Hz stimulation (180deg phase lag between both sites). To ensure a consistent phase lag, stimulation will be applied for 1min, then stopped and restarted after 5s. The sham stimulation will make use of vibrations at 6Hz instead of electrical current to mimic the physical throbbing sensation.

ELIGIBILITY:
Inclusion Criteria:

* Right-handedness
* Normal cognitive functions (>25 on Montreal Cognitive Assessment Questionnaire)
* Normal vision
* Healthy

Exclusion Criteria:

* Transcranial Electric Stimulation (TES) is contra-indicated (TES screening questionnaire)
* Neurologic or psychiatric disorders
* Physical disorder(s) that might interfere with the execution of the bimanual motor task
* Alcohol and/or drug addiction
* Active smokers
* Current use of specific drugs that interfere with the central nervous system
* Skin allergies to cosmetics and lotions
* Pregnancy

Ages: 65 Years to 77 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Bimanual Coordination accuracy during the stimulation or sham | day 1
  This is a motor performance measure on the bimanual tracking task that will be used in this project. The measure combines the average distance of the subject's cursor to the requested target's position, and the Euclidean distance of the subject's cursor position to the target line that has to be followed. This will be measured in the blocks that were executed during the (sham) stimulation.
Bimanual Coordination accuracy during the stimulation or sham | day 25
  This is a motor performance measure on the bimanual tracking task that will be used in this project. The measure combines the average distance of the subject's cursor to the requested target's position, and the Euclidean distance of the subject's cursor position to the target line that has to be followed. This will be measured in the blocks that were executed during the (sham) stimulation.
Bimanual Coordination accuracy during the stimulation or sham | day 49
  This is a motor performance measure on the bimanual tracking task that will be used in this project. The measure combines the average distance of the subject's cursor to the requested target's position, and the Euclidean distance of the subject's cursor position to the target line that has to be followed. This will be measured in the blocks that were executed during the (sham) stimulation.
Bimanual Coordination accuracy 15 minutes after stimulation or sham | day 1
  This is a motor performance measure on the bimanual tracking task that will be used in this project. The measure combines the average distance of the subject's cursor to the requested target's position, and the Euclidean distance of the subject's cursor position to the target line that has to be followed. This will be measured in the retention block that was executed 15min after the (sham) stimulation.
Bimanual Coordination accuracy 15 minutes after stimulation or sham | day 25
  This is a motor performance measure on the bimanual tracking task that will be used in this project. The measure combines the average distance of the subject's cursor to the requested target's position, and the Euclidean distance of the subject's cursor position to the target line that has to be followed. This will be measured in the retention block that was executed 15min after the (sham) stimulation.
Bimanual Coordination accuracy 15 minutes after stimulation or sham | day 49
  This is a motor performance measure on the bimanual tracking task that will be used in this project. The measure combines the average distance of the subject's cursor to the requested target's position, and the Euclidean distance of the subject's cursor position to the target line that has to be followed. This will be measured in the retention block that was executed 15min after the (sham) stimulation.
Stability of movement during the stimulation or sham | day 1
  This is a motor performance measure on the bimanual tracking task that will be used in this project. This measure is calculated by fitting a straight line through the participant's own trajectory and then measuring the average Euclidean distance of the subject's cursor position to the fitted line of the trajectory. This will be measured in the blocks that were executed during the (sham) stimulation.
Stability of movement during the stimulation or sham | day 25
  This is a motor performance measure on the bimanual tracking task that will be used in this project. This measure is calculated by fitting a straight line through the participant's own trajectory and then measuring the average Euclidean distance of the subject's cursor position to the fitted line of the trajectory. This will be measured in the blocks that were executed during the (sham) stimulation.
Stability of movement during the stimulation or sham | day 49
  This is a motor performance measure on the bimanual tracking task that will be used in this project. This measure is calculated by fitting a straight line through the participant's own trajectory and then measuring the average Euclidean distance of the subject's cursor position to the fitted line of the trajectory. This will be measured in the blocks that were executed during the (sham) stimulation.
Stability of movement 15 minutes after the stimulation or sham | day 1
  This is a motor performance measure on the bimanual tracking task that will be used in this project. This measure is calculated by fitting a straight line through the participant's own trajectory and then measuring the average Euclidean distance of the subject's cursor position to the fitted line of the trajectory. This will be measured in the retention block that was executed 15min after the (sham) stimulation.
Stability of movement 15 minutes after the stimulation or sham | day 25
  This is a motor performance measure on the bimanual tracking task that will be used in this project. This measure is calculated by fitting a straight line through the participant's own trajectory and then measuring the average Euclidean distance of the subject's cursor position to the fitted line of the trajectory. This will be measured in the retention block that was executed 15min after the (sham) stimulation.
Stability of movement 15 minutes after the stimulation or sham | day 49
  This is a motor performance measure on the bimanual tracking task that will be used in this project. This measure is calculated by fitting a straight line through the participant's own trajectory and then measuring the average Euclidean distance of the subject's cursor position to the fitted line of the trajectory. This will be measured in the retention block that was executed 15min after the (sham) stimulation.
Working Memory during stimulation or sham | Day 1
  Working memory will be assessed using the sensitivity index. This will be measured in the blocks that were executed during the (sham) stimulation.
Working Memory during stimulation or sham | Day 25
  Working memory will be assessed using the sensitivity index. This will be measured in the blocks that were executed during the (sham) stimulation.
Working Memory during stimulation or sham | Day 49
  Working memory will be assessed using the sensitivity index. This will be measured in the blocks that were executed during the (sham) stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Bart Van Wijmeersch, prof. dr., Study Director — Hasselt University; Raf Meesen, prof. dr., Principal Investigator — Hasselt University; Stefanie Verstraelen, drs., Study Chair — Hasselt University; Kim van Dun, dr., Study Chair — Hasselt University
Locations (1):
- Hasselt University, Hasselt, Belgium

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers